CLINICAL TRIAL: NCT04918433
Title: Comparison of Pectointercostal Block and Transverse Thoracic Plane Block for ERAS Post Congenital Cardiac Surgery
Brief Title: Comparison of Two Regional Anaesthetic Blocks for ERAS After Congenital Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Ibrahim Mabrouk Ibrahim, Assistant lecturer, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Local Infiltration
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRANSEVERSUS THORACIS MUSCLE PLANE BLOCK (TTPB) (Active Comparator): After induction of anaesthesia, ultrasound guided transverses thoracis muscle plane block will be done using 0.25% bupivacaine
  Interventions: Procedure: Regional anaesthesia
- PECTO-INTERCOSTAL FACIAL PLANE BLOCK (PIFB) (Active Comparator): After induction of anaesthesia, ultrasound guided pectointercostal facial plane block will be done using 0.25% bupivacaine
  Interventions: Procedure: Regional anaesthesia

INTERVENTIONS:
Procedure: Regional anaesthesia — Regional anaesthesia for sternotomy incision for congenital cardiac surgery

SUMMARY:
The current study is designed to compare the perioperative analgesic efficacy of transversus thoracis plane block (TTPB) and Pecto-intercostal-fascial plane block (PIFB) in children undergoing cardiac surgery via median sternotomy

DETAILED DESCRIPTION:
Sixty paediatric patients of either sex, aged 2-12 years, undergoing elective cardiac surgery via median sternotomy. Patients will be excluded from the current study in case of, refusal to participate, redo or urgent cardiac surgery, local infection of the skin at the site of needle puncture, allergy to bupivacaine, coagulation disorders, clinically significant liver or kidney disease, heart failure, moderate to severe pulmonary hypertension, and when extubation is intentionally planned to be delayed. Patients will be randomly assigned to one of two equal groups, the PIF block group and TTP block group, each will include 30 patients, by a computer-generated randomization table and concealed sealed opaque envelopes.

ELIGIBILITY:
Inclusion Criteria:

* either sex, aged 2-12 years, undergoing

elective cardiac surgery via median sternotomy

Exclusion Criteria:

* refusal to participate, redo or urgent cardiac surgery, local infection of the skin at the site of needle puncture, allergy to bupivacaine, coagulation disorders, clinically significant liver or kidney disease, heart failure, moderate to severe pulmonary hypertension

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
Weight, height , BMI | 1 year
  Weight in kg and height in cm to allow BMI measurement weight (kg) / height (m2)
Postoperative pain score | 1 year
  Postoperative pain score at rest, hemodynamic effects, analgesic consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No